CLINICAL TRIAL: NCT04671433
Title: Phase 3 Randomized, Controlled Study of AAV5-hRKp.RPGR for the Treatment of X-linked Retinitis Pigmentosa Associated With Variants in the RPGR Gene
Brief Title: Gene Therapy Trial for the Treatment of X-linked Retinitis Pigmentosa Associated With Variants in the RPGR Gene
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR109258; MGT-RPGR-021 (Other: Janssen Research & Development, LLC); 2020-002873-88 (EudraCT Number)
Record Dates: First submitted 2020-11-05; First posted 2020-12-17 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: X-Linked Retinitis Pigmentosa

STUDY DESIGN:
Intervention Model Description: Bilateral, subretinal administration of AAV5-RPGR - immediate treatment group
Who Masked: Outcomes Assessor
Masking Description: No intervention - deferred treatment group (Bilateral, subretinal administration of AAV5-RPGR to be administered in the follow-up study)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Experimental - Immediate Treatment (Experimental): Intermediate dose.
  Interventions: Biological: Genetic: AAV5-hRKp.RPGR
- Deferred Treatment (Other): Deferred Treatment
  Interventions: Biological: Genetic: AAV5-hRKp.RPGR
- Experimental Immediate Treatment (Experimental): Low dose.
  Interventions: Biological: Genetic: AAV5-hRKp.RPGR

INTERVENTIONS:
Biological: Genetic: AAV5-hRKp.RPGR — Bilateral, sub-retinal administration of AAV5-hRKp.RPGR - immediate treatment group
  Other Names: botaretigene sparoparvovec
  Arms: Experimental - Immediate Treatment; Experimental Immediate Treatment
Biological: Genetic: AAV5-hRKp.RPGR — No intervention - deferred treatment group (Bilateral, sub-retinal administration of AAV5-hRKp.RPGR to be administered in the follow-up study)
  Arms: Deferred Treatment

SUMMARY:
A clinical trial of AAV5-RPGR vector for participants with X-linked retinitis pigmentosa (XLRP)

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 3 years of age or older
* Has XLRP confirmed by a retinal specialist and has a predicted disease-causing sequence variant in RPGR confirmed by an accredited laboratory

Exclusion Criteria:

* Has had ocular surgery within 3 months prior to screening or is anticipated to require ocular surgery within 6 months after the study intervention administration
* Any investigational ocular treatment or any other ocular treatment that could confound the interpretation of the efficacy results or affect participant compliance with the visit schedule
* Has undergone prior retinal surgery involving the macula, macular laser photocoagulation, external-beam radiation therapy, transpupillary thermotherapy, glaucoma filtration surgery or corneal surgery

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change From Baseline to Week 52 in Vision-guided Mobility Assessment (VMA) as Measured by the Ability of the Participant to Navigate Through a VMA Maze | From Baseline to 52 Weeks
  Change from baseline to Week 52 in VMA as measured by the ability of the participant to navigate through a VMA maze.

SECONDARY OUTCOMES:
Change From Baseline in Mean Retinal Sensitivity Within the Central 10 Degrees Excluding Scotoma (Mean Retinal Sensitivity Within the Central 10 Degree Excluding Scotoma in Static Perimetry [MRS10]) in Static Perimetry at Week 52 | From Baseline to Week 52
  Change from baseline in mean retinal sensitivity within the central 10 degrees excluding scotoma (MRS10) in static perimetry at Week 52 will be assessed.
Change From Baseline in Mean Retinal Sensitivity of Worse-seeing Eye Within the Central 10 Degrees Excluding Scotoma in Static Perimetry (MRS10) at Week 52 | From Baseline to Week 52
  Change from baseline in mean retinal sensitivity of worse-seeing eye within the central 10 degrees excluding scotoma in static perimetry (MRS10) at Week 52 will be assessed.
Change in Retinal Function as Assessed by Pointwise Response in Full Visual Field at Week 52 | From Baseline to Week 52
  Pointwise response in full visual field at Week 52 will be assessed.
Change in Retinal Function as Assessed by Pointwise Response in Worse-seeing Eye in Full Visual Field at Week 52 | From Baseline to Week 52
  Pointwise response in worse-seeing eye in full visual field at Week 52 will be assessed.
Change in Retinal Function as Assessed by Pointwise Response in the Central 30 Degrees Visual Field at Week 52 | From Baseline to Week 52
  Pointwise response in the central 30 degrees visual field at Week 52 will be assessed.
Change in Retinal Function as Assessed by Pointwise Response in Worse-seeing Eye in the Central 30 Degrees Visual Field at Week 52 | From Baseline to Week 52
  Pointwise response in worse-seeing eye in the central 30 degrees visual field at Week 52 will be assessed.
Change From Baseline in Retinal Function as Assessed by Mean Retinal Sensitivity Within the Full Visual Field (MRS90) in Static Perimetry at Week 52 | From Baseline to Week 52
  Change from baseline in retinal function as assessed by mean retinal sensitivity within the full visual field (MRS90) in static perimetry at Week 52 will be assessed.
Change in Functional Vision by Using Vision-guided Mobility Assessment (VMA) Response in the "Worse-seeing Eye" at Week 52 | From Baseline to Week 52
  Change in functional vision by using VMA assessment in the "Worse-seeing Eye" at Week 52.
Change From Baseline in the Modified Low Luminance Questionnaire (mLLQ) Extreme Lighting Domain score at Week 52 | From Baseline to Week 52
  Change From Baseline in the Modified Low Luminance Questionnaire (mLLQ) Extreme Lighting Domain score at Week 52.
Change From Baseline in Visual Function as Assessed by Monocular Low Luminance Visual Acuity Using the Early Treatment Diabetic Retinopathy Study (ETDRS) Chart Letter score at Week 52 | From Baseline to Week 52
  Change from baseline in visual function as assessed by monocular low luminance visual acuity using the ETDRS chart letter score at Week 52.
Change From Baseline in Visual Function as Assessed by monocular Best Corrected Visual Acuity (BCVA) Using the ETDRS Chart Letter Score at Week 52 | From Baseline to Week 52
  Change From Baseline in visual function as assessed by monocular BCVA using the ETDRS chart letter score at Week 52.
Change From Baseline in Visual Function as Assessed by Low Luminance Visual Acuity Using the ETDRS Chart Letter Score in Worse-seeing Eye at Week 52 | From Baseline to Week 52
  Change from baseline in visual function as assessed by low luminance visual acuity using the ETDRS chart letter score in worse-seeing eye at Week 52.
Number of Participants with Ocular and Non-ocular Adverse Events | Day 1 - Week 52
  Number of participants with ocular and non-ocular adverse events will be assessed.
Number of Participants With Abnormalities in Laboratory Assessments | Day 1 - 52 Weeks
  Number of participants with abnormalities in laboratory assessments will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (27):
- United States (9):
  - Shiley Eye Institute Jacobs Retina Center, La Jolla, California
  - Childrens Hospital, Los Angeles, California
  - Stanford Health Care, Palo Alto, California
  - VitreoRetinal Associates, PA, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital - Center for Celiac Research and Treatment, Boston, Massachusetts
  - Univ of Michigan Medical Center, Ann Arbor, Michigan
  - Duke Eye Center, Durham, North Carolina
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
- UZ Gent, Ghent, Belgium
- Hospital For Sick Children, Toronto, Ontario, Canada
- Rigshospitalet Glostrup, Glostrup Municipality, Denmark
- Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts, Paris, France
- Hadassah Medical Center, Jerusalem, Israel
- Italy (4):
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Ospedale San Paolo, Milan
  - Azienda Ospedaliera Univ.- Università Degli studi della Campania - Luigi Vanvitelli, Napoli
  - IRCCS Fondazione G.B. Bietti per lo Studio e la Ricerca in Oftalmologia ONLUS, Roma
- Netherlands (2):
  - VUMC Amsterdam, Amsterdam
  - Radboudumc, Nijmegen
- Hosp Univ Fund Jimenez Diaz, Madrid, Spain
- Switzerland (2):
  - University Hospital Basel, Eye Clinic/Institute of Molecular and Clinical, Basel
  - Universite de Lausanne, Hopital ophtalmique Jules-Gonin, Lausanne
- United Kingdom (4):
  - NHS Lothian, Edinburgh
  - Gartnavel General Hospital, Glasgow
  - St James University Hospital, Leeds
  - Moorfields Eye Hospital, London

IPD SHARING:
Plan to Share IPD: No